CLINICAL TRIAL: NCT02706093
Title: Metabolic Adaptations in Response to High Intensity Interval Training in Obese Adults
Acronym: HT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jeffrey F Horowitz, Professor, Movement Science and Director, Substrate Metabolism Laboratory, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HUM00106883
Record Dates: First submitted 2016-03-02; First posted 2016-03-11 (Estimated); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Glucose Intolerance
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- High Intensity Interval Training #1 (Other): Obese adults with impaired glucose tolerance will be randomized into one of four different exercise training groups for a 3 month exercise intervention.
  Interventions: Other: High Intensity Interval Training #1
- Moderate intensity continuous training (Other): Obese adults with impaired glucose tolerance will be randomized into one of four different exercise training groups for a 3 month exercise intervention.
  Interventions: Other: Moderate intensity continuous training
- High Intensity Interval Training #2 (Other): Obese adults with impaired glucose tolerance will be randomized into one of four different exercise training groups for a 3 month exercise intervention.
  Interventions: Other: High Intensity Interval Training #2
- High Intensity Interval Training #3 (Other): Obese adults with impaired glucose tolerance will be randomized into one of four different exercise training groups for a 3 month exercise intervention.
  Interventions: Other: High Intensity Interval Training #3

INTERVENTIONS:
Other: High Intensity Interval Training #1 — (HIIT#1) 10 x 1 min. at ~90%HRmax - with low intensity warm-up, recovery, and cool down - total of 25 min/session .
  Arms: High Intensity Interval Training #1
Other: Moderate intensity continuous training — Moderate-intensity continuous training (MICT) = steady-state exercise at 60-70%HRmax for 45min. Representing a commonly prescribed exercise program.
  Arms: Moderate intensity continuous training
Other: High Intensity Interval Training #2 — (HIIT #2) 5 x 1 min at 90%HRmax + 10 min steady-state exercise at 70%HRmax [25min; ~150kcals; 4d/wk]
  Arms: High Intensity Interval Training #2
Other: High Intensity Interval Training #3 — (HIIT #3) 5 x 1 min at 90%HRmax [15min; ~90kcals; 4d/wk]
  Arms: High Intensity Interval Training #3

SUMMARY:
The overall objectives are to:

1. Assess mechanisms underlying HIIT-induced improvements in insulin resistance at the whole-body, tissue, and cellular levels.
2. Systematically compare different HIIT regimens to help identify effective "doses" of HIIT that may be optimal for improving metabolic health in obese adults.
3. Assess the ability/willingness of obese subjects to adhere to a long-term HIIT program.

Findings from these studies will greatly expand knowledge about the effects of HIIT on metabolic health, and will provide valuable information for development of programs aimed at maximizing key metabolic benefits of exercise.

DETAILED DESCRIPTION:
If subjects are eligible for the study, they will be randomized into one of four different exercise training groups. Before training (and twice after 3 months of training) subjects will participate in a "clinical study" in which they will be required to stay overnight in the hospital. During the clinical study, the research team will perform a series of metabolic tests. Before and after the 3 months of training, the research team will assess subjects "free-living" 24h blood sugar control using a Continuous Glucose Monitor (CGM). The research team will measure several other relevant clinical markers (e.g., whole body and regional body fat assessments [Dual Energy X-ray Absorptiometry (DEXA) and Magnetic Resonance Imager (MRI)], hepatic lipid accumulation [MRI analysis], blood lipid profile, resting metabolic rate, glycated hemoglobin [hemoglobin A1c]). After the first 3 months of training, adherence to the subjects assigned training program will be tracked for the next 9 months (1 year of training in total). One year after initiating a training program, subjects will be asked to return to the clinic for a quick follow-up visit where the research team will complete some standard clinical assessments (e.g., body weight, body composition, blood pressure, and a blood sample).

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-40
* Body Mass Index: 30-40 kg/m2
* Waist circumference: 88-98cm for women and 100-110cm for men
* Glucose intolerant (i.e., 2h glucose concentration during a screening oral glucose tolerance test (OGTT)= 140-199mg/dl
* No regularly planned exercise/physical activity
* Women must have regularly occurring menses and must be premenopausal

Exclusion Criteria:

* EKG abnormalities as assessed by the cardiologist on the research team
* Evidence/history of cardiovascular or metabolic disease
* Medications known to affect lipid or glucose metabolism
* Pregnant or lactating
* Tobacco or e-cigarette use

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 129 (Actual)
Dates: Start 2016-05-03 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-05-04 (Actual)

PRIMARY OUTCOMES:
Insulin Sensitivity | Change from Baseline at 3 months
  A hyperinsulinemic-euglycemic clamp will be used to assess peripheral insulin sensitivity

SECONDARY OUTCOMES:
Continuous Glucose Monitoring | Change from Baseline at 3 months
Resting Metabolic Rate | baseline and 3 months
Muscle Biopsy | Change from Baseline at 3 months
  To measure Mitochondrial Proteins
Adipose Tissue Biopsy | Change from Baseline at 3 months
  To measure cytokines

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Horowitz, Principal Investigator — University of Michigan
Locations (1):
- Suzette Howton, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ryan BJ, Schleh MW, Ahn C, Ludzki AC, Gillen JB, Varshney P, Van Pelt DW, Pitchford LM, Chenevert TL, Gioscia-Ryan RA, Howton SM, Rode T, Hummel SL, Burant CF, Little JP, Horowitz JF. Moderate-Intensity Exercise and High-Intensity Interval Training Affect Insulin Sensitivity Similarly in Obese Adults. J Clin Endocrinol Metab. 2020 Aug 1;105(8):e2941-59. doi: 10.1210/clinem/dgaa345. PMID 32492705